CLINICAL TRIAL: NCT05064423
Title: Clinical Trials Outreach & Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MCC-21235; 3P30CA076292-21S3 (NIH)
Record Dates: First submitted 2021-09-22; First posted 2021-10-01 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Knowledge, Attitudes, Practice
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Trials Education (Experimental): Community Health Educators (CHE) will provide Clinical Trial Education to increase knowledge of Clinical Trials and the importance of Clinical Trial participation.
  Interventions: Behavioral: Clinical Trials Education Program

INTERVENTIONS:
Behavioral: Clinical Trials Education Program — The Community Health Educator (CHE) will provide CT education and outreach to increase clinical trial knowledge and the importance of clinical trials research and participation. The clinical trials educational activities will include the use of NCI Colorectal Cancer resources and materials, including a PowerPoint presentation, clinical trials information, and online resources. The CHE will tailor the PowerPoint slides to ensure that they are culturally tailored, visually appealing, low-literacy, language appropriate and include appropriate visuals. The CTs educational sessions will be delivered in Spanish and English and will take approximately 45 minutes to 1 hour.

SUMMARY:
The purpose of this study is to provide education and information about clinical trials and clinical trials participation. Investigators also aim to see if education makes a difference in increasing knowledge of clinical trials and clinical trials participation.

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* Able to provide informed consent
* Reside in the Tampa Bay Area (Hillsborough, Pinellas, Polk or Pasco county)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-23 (Actual); Study Completion 2022-03-23 (Actual)

PRIMARY OUTCOMES:
Change in Participants Clinical Trials Knowledge | Change from baseline to immediately after receiving intervention
  To assess the impact of the educational intervention on participants knowledge and beliefs about clinical trials, participants will be asked to complete a survey prior to and after the educational intervention. The pre-assessment and post assessment survey includes 11 items assessing knowledge of clinical trials, risks and benefits to clinical trials participation, and the consent process. Additionally, the assessment includes 6 items to determine intentions to seek out information related to clinical trials, speak with one's healthcare provider about appropriate clinical trials, clinical trials participation, and talking with family/friends about participating in clinical trials.

CONTACTS AND LOCATIONS:
Overall Officials: Clement K Gwede, PhD, MPH, RN, FAAN, Principal Investigator — Moffitt Cancer Center
Locations (1):
- Moffitt Cancer Center, Tampa, Florida, United States